CLINICAL TRIAL: NCT01589523
Title: Conjugated Cholic Acid for the Treatment of Inborn Errors in Bile Acid Synthesis Involving Side-Chain Conjugation
Brief Title: GlycoCholic Acid Treatment for Patients With Inborn Errors in Bile Acid Synthesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0780
Record Dates: First submitted 2012-04-03; First posted 2012-05-02 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Bile Acid Synthesis Defect; Inborn Error of Bile Acid Metabolism; Inborn Error of Bile Acid Conjugation
MeSH Terms: interventions — Glycocholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GlycoCholic Acid, Study Drug (Experimental): An open label, single arm, non-randomized, non-comparative, treatment study of Glycocholic Acid in the treatment of defects of bile acid metabolism.
  Interventions: Drug: Glycocholic Acid

INTERVENTIONS:
Drug: Glycocholic Acid — 10-15mg/kg body weight/day taken orally. Supplied as either liquid or 50mg capsules.
  Other Names: Conjugated Cholic Acid

SUMMARY:
The purpose of this research study is to determine the way (mechanisms) by which your defect in bile acid handling (metabolism) causes your liver disease or abnormality in absorption of vitamins and the effect of an investigational bile acid therapy (glycocholic acid) on your vitamin absorption and your liver disease. An investigational therapy is one that not approved by the United States Food and Drug Administration (FDA) and is being provided to you under an Investigational New Drug application from the FDA.

DETAILED DESCRIPTION:
Inborn errors of bile acid metabolism have been established as a well recognized cause of neonatal cholestasis and fat-soluble vitamin malabsorption. Although there is extensive experience with metabolic defects in the biosynthetic pathway, few patients have identified with defects in conjugation with taurine or glycine that allows bile acids to become effective detergents. This protocol is designed to study the effect of defects of conjugation of bile acids on growth and fat-soluble vitamin malabsorption. Study subjects will have liver function studies performed, serum and urinary bile acid measurements, vitamin levels, growth measurements, bile acid pool size measurements made by stable isotope dilution mass-spectrometry, and measurements of absorption of two fat-soluble vitamins, tocopherol and vitamin D. Subjects will be treated orally with conjugates of cholic acid with follow-up laboratories performed as an outpatient and then subjects will have all of the initial studies repeated during an inpatient stay 3-12 months after starting treatment. Subjects with previous liver biopsies indicating the presence of significant liver disease will have a repeat liver biopsy after 3-12 months treatment to assess the histologic response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of a diagnosis of an inborn error of bile acid synthesis/conjugation based upon urine analysis by FAB-MS.
2. Any age
3. Participant must be willing and able to comply with study assessments and procedures.
4. The participant and/or parent/legal guardian must have signed the written informed consent document prior to study start.

Exclusion Criteria

1. No confirmed diagnosis of inborn error of bile acid synthesis/conjugation based upon urine analysis by FAB-MS.

Ages: 1 Week to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-02; Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D. Setchell, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; James E. Heubi, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Setchell KD, Heubi JE, Shah S, Lavine JE, Suskind D, Al-Edreesi M, Potter C, Russell DW, O'Connell NC, Wolfe B, Jha P, Zhang W, Bove KE, Knisely AS, Hofmann AF, Rosenthal P, Bull LN. Genetic defects in bile acid conjugation cause fat-soluble vitamin deficiency. Gastroenterology. 2013 May;144(5):945-955.e6; quiz e14-5. doi: 10.1053/j.gastro.2013.02.004. Epub 2013 Feb 13. PMID 23415802
- [Result] Heubi JE, Setchell KD, Jha P, Buckley D, Zhang W, Rosenthal P, Potter C, Horslen S, Suskind D. Treatment of bile acid amidation defects with glycocholic acid. Hepatology. 2015 Jan;61(1):268-74. doi: 10.1002/hep.27401. Epub 2014 Dec 23. PMID 25163551

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycocholic Acid: 15 milligrams/kilograms (mg/kg) of body weight/day (bw/day)
Period: Overall Study
Arm/Group | Glycocholic Acid
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glycocholic Acid
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Conjugated Cholic Acid (GCA) for the Treatment of Inborn Errors in Bile Acid Synthesis Involving Side-chain Conjugation.
Description: This is the number of participants with bile acid amidation defects treated with oral glycocholic acid (15 milligrams/kilograms (mg/kg) of body weight/day (bw/day))
Time Frame: Up to 10 years
Measure: Count of Participants; unit: Participants
Groups:
- 15 mg/Kg Body Weight/Day: Open-label, no placebo group. Participants with bile acid conjugation defect confirmed by urine mass spectrometry analysis receiving glycocholic acid (15 mg/kg bw/day)
Arm/Group | 15 mg/Kg Body Weight/Day
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Evaluation of Levels of Atypical Bile Acid Metabolites After GCA Treatment Compared
Description: Semi-quantitative descriptive evaluation of the levels of atypical bile acids in urine measured by mass spectrometry (FAB MS) based on a scale of 0 = absent or traces levels, 1 = low levels, 2 = moderate levels, 3 = high levels using the signal/noise ratio and intensity of ions. Atypical bile acids evaluated included m/z 407 (unconjugated cholic acid), m/z 471 (dihydroxy-choleanoic-sulfate) and m/z 583 (trihydroxy-choleanoic glucuronide).
Time Frame: Average of 6 months, average 12 months, and average of after year 1 to 10 years
Measure: Median (Full Range); unit: score on a scale
Groups:
- 10-15 mg/Kg Body Weight/Day: Open-label, no placebo group. Participants with bile acid conjugation defect confirmed by urine mass spectrometry analysis receiving glycocholic acid (10-15 mg/kg bw/day)
Arm/Group | 10-15 mg/Kg Body Weight/Day
Number analyzed (Participants) | 5
score on a scale
  6 months average: number analyzed (Participants) | 2
  6 months average | 1.4 [0 to 2.0]
  12 months average: number analyzed (Participants) | 2
  12 months average | 1 [1 to 1]
  average of year 1 to 10 | 1 [0 to 3]

3. Secondary Outcome: Changes in Liver Function Tests of ALT From Baseline to Post-treatment
Description: Liver function tests Alanine Aminotransferease (ALT)
Time Frame: Comparison between baseline and post-treatment (average of available timepoints after year 1 through year 10)
Measure: Mean (Standard Error); unit: units per liter (U/L)
Arm/Group | Glycocholic Acid
Number analyzed (Participants) | 5
units per liter (U/L)
  Baseline | 43.8 (10.5)
  average of available timepoints after year 1 through year 10 | 31.7 (2.2)
Statistical Analysis 1: Comparison: Glycocholic Acid; Test type: Equivalence — paired t-test; p = 0.342, t-test, 2 sided

4. Secondary Outcome: Change in Liver Function Test: AST From Baseline to Post-treatment
Description: Measure of Aspartate Aminotransferase (AST)
Time Frame: Comparison between baseline and post-treatment (average of available timepoints after year 1 through year 10)
Measure: Median (Standard Error); unit: units per liter (U/L)
Arm/Group | Glycocholic Acid
Number analyzed (Participants) | 4
units per liter (U/L)
  Baseline | 65 (14.2)
  average of available timepoints after year 1 through year 10 | 39 (3.5)
Statistical Analysis 1: Comparison: Glycocholic Acid; Test type: Equivalence — paired t-test; p = 0.116, t-test, 2 sided

5. Secondary Outcome: Change in Vitamin D, 25-OH Measure From Baseline to Post-treatment
Description: Measure Vitamin D levels nanograms per milliliter (ng/mL)
Time Frame: Pre-treatment and post treatment (average of available timepoints after year 1 through year 10)
Population: Missing data on Vitamin D from 2 participants.
Measure: Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | Glycocholic Acid
Number analyzed (Participants) | 3
nanograms per milliliter (ng/mL)
  Baseline | 1.0 (0.8)
  average of available timepoints after year 1 through year 10 | 25.7 (5.9)
Statistical Analysis 1: Comparison: Glycocholic Acid; Test type: Equivalence — paired t-test; p = 0.065, t-test, 2 sided; vitamin D

ADVERSE EVENTS:
Time Frame: Adverse events were assessed while patients were receiving investigational agent; up to 10 years.
Groups:
- Glycocholic Acid: 15 mg/kg bw/day
Arm/Group | Glycocholic Acid
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT01589523/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT01589523/ICF_001.pdf